CLINICAL TRIAL: NCT05225987
Title: The Effect of Nurse Navigation Program Developed for Postpartum Mothers on Mothers' Self-Care Power, Quality of Life, Anxiety and Depression Risks, and Physical Symptom Severity
Brief Title: Effects of Postpartum Nurse Navigation Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pinar Uzunkaya Oztoprak, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020/12
Record Dates: First submitted 2021-06-11; First posted 2022-02-07 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Nursing Caries; Nurse's Role; Postpartum Depression; Postpartum Anxiety; Quality of Life; Postpartum Disorder
Keywords: Postpartum; Nurse Navigation Program; Quality of life; Self care power; Postpartum depression
MeSH Terms: conditions — Depression, Postpartum; Puerperal Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal Group (Experimental): Postpartum Nurse Navigation Program based care
  Interventions: Behavioral: Postpartum Nurse Navigation Program based care
- Control group (No Intervention): This group will take routin care

INTERVENTIONS:
Behavioral: Postpartum Nurse Navigation Program based care — In addition to routine hospital care, the intervention group will receive navigation program-based nursing care that includes three home visits, three phone calls, and sending text messages at five different times.
  Arms: Experimantal Group

SUMMARY:
The study was planned as a two-group parallel randomized controlled experimental study in order to determine the effects of the nurse navigation program developed for mothers in the postpartum period on mothers' self-care power, quality of life, anxiety and depression risks, and physical symptom severity. The study will be carried out in Ankara Etlik Zübeyde Hanım Gynecology Training and Research Hospital. The population of the research will be primiparous mothers who gave birth vaginally in Ankara.

DETAILED DESCRIPTION:
Primiparous pregnant women who come to the pregnancy outpatient clinic, are at 36 weeks of gestation or more, meet the inclusion criteria and volunteer, will be informed about the program and will be included in the sample of the study. There will be two groups assigned by the stratified block randomization method in the study. The number of samples to be taken into the control and intervention groups was determined by power analysis and the sample size was planned to be 32 mothers for the intervention group and 32 mothers for the control group. In addition to routine hospital care, the intervention group will receive navigation program-based nursing care that includes three home visits, three phone calls, and sending text messages at five different times. The control group will not receive any intervention other than routine hospital care practices. The data of the research; "Data Collection Form on Descriptive Characteristics", "Postpartum Mother and Newborn Evaluation and Diagnosis Form", "Mother and Newborn Problems Evaluation Form in the Postpartum Period", "Mother and Baby Follow-up Evaluation Form in the Postpartum Period", "Self-Care Power" Scale', 'Postpartum Quality of Life Scale', 'Postpartum Specific Anxiety Scale', 'Edinburgh Postpartum Depression Scale' and 'Physical Symptom Severity Scale' will be collected using descriptive statistics (number, min., mean, standard deviation, standard deviation) in the evaluation of the data. max.) will be used. The conformity of the data to the normal distribution will be evaluated with the Shapiro Wilks test. The relationship between them in qualitative variables will be evaluated with the chi-square test and Fisher's exact test. The Cochran Q test will be used to examine change over time. In numerical variables, according to the normal distribution; In independent groups, t test, Mann Whitney U test, one-way analysis of variance (ANOVA), Kruskal Wallis Analysis will be used. Before and after repeated measurements, according to the normal distribution; In repeated measurements, one-way analysis of variance or Friedman test will be used. Significance will be evaluated at the p<0.05 level. The independent variables of the research will be stated as numbers and percentages.

ELIGIBILITY:
Inclusion Criteria:

1. between the ages of 18-45
2. gestational week ≥36,
3. primiparous and singleton pregnancy,
4. no vision and hearing problems,
5. able to communicate via telephone,
6. no complications during pregnancy and delivery (preeclampsia; eclapsia; diabetes; 7. hypertension; heart disease; kidney failure; HIV /AIDS)

8. pregnant women will be included.

Exclusion Criteria:

1. Mothers who were illiterate,
2. had problems in communicating,
3. did not have a mobile phone of their own,
4. residing outside the province of Ankara,
5. had mental disability and severe mental illness and
6. had preterm or postterm birth will exclude from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Self-Care Power Scale Score | 5 months
  The Self-Care Power Scale was developed by Kearney and Fleischer (1979) to determine individuals' ability to take care of themselves. Its Turkish validity and reliability was determined by Nahçıvan (1993), and the Cronbach α coefficient of the scale was stated as 0.89 (Nahcivan, 2004).
  The Scale consists of 35 items. Each item of this 5-point Likert-type scale, according to the answer given; It is evaluated by giving 0 points for the answer "Doesn't describe me at all", and 4 points for the answer "It describes me a lot". Evaluation is made out of a total of 140 points. Below 82 points is considered as low, 82-120 points as medium, above 120 points as high (Nahcivan, 2004).
Postpartum Quality of Life Scale Score | 5 months
  It was developed by Hill et al (2006) to evaluate the postpartum quality of life of mothers. The Turkish validity and reliability study of the scale was carried out by Altuntuğ and Ege (2012), and the internal consistency coefficient of the scale was determined as 0.95 in the study (Altuntuğ & Ege, 2012).
  In the first part of the scale, satisfaction with each item is questioned, and in the second part, the importance is questioned. All items are evaluated on a 6-point Likert scale. Satisfaction and Significance sections of the scale are numbered from 1 to 6. 1=Not at all Satisfied, 2=Moderately Dissatisfied, 3=Slightly Dissatisfied, 4=Slightly Satisfied, 5=Moderately Satisfied, 6=Very Satisfied. The Quality of Life Score is in the range of 0-30. The higher the score obtained from the scale, the higher the person's postpartum quality of life, and lower scores the lower the postpartum quality of life (Hill et al. 2006, Altuntuğ & Ege, 2012).
Postpartum Specific Anxiety Scale Score | 5 months
  Fallon et al. (2016) to evaluate postpartum anxiety symptoms (Fallon et al, 2016). The Turkish validity and reliability study of the scale was conducted by Duran (2019), and the internal consistency coefficient of the scale was determined as 0.91 in the study (Duran, 2019).
  The scale consists of 51 items. It has been stated that those who score 73 and below on the scale have low postpartum anxiety levels, those who score between 74 and 100 have a medium level, and those who score 101 and above have a high level (Duran, 2019). The scale was administered within 6 months of postpartum and it was recommended to be used during this period. In the development of the scale, retests were performed 2 weeks after the scale was applied (Fallon et al, 2016).
Edinburgh Postpartum Depression Scale Score | 5 months
  It was developed by Cox (1987). The scale is a self-report scale aimed at screening postpartum depression in women (Cox et al, 1987). The Turkish validity and reliability study of the scale was carried out by Engindeniz et al. (1996), and they found the internal consistency coefficient of the scale as 0.79 (Engindeniz et al., 1996). In this study, the Cronbach α value of the scale will be calculated.
  EPDS consists of 10 items. Each item of the scale is evaluated in a 4-point Likert format and the answer given to each item is scored between 0 and 3 (0, 1, 2, 3). The lowest score that can be obtained from the scale is 0, and the highest score is 30. In the evaluation of the scale, the 1st, 2nd and 4th items are scored as 0-1-2-3, while the 3rd, 5th, 6th, 7th, 8th, 9th and 10th items are scored as 3-2-1-0. are scored inversely. The cut-off point of the scale is 12. Women with a score of 12 and above are considered to be at risk for depression (Engindeniz, 1996).
Physical Symptom Severity Scale Score | 5 months
  The scale was developed by Cine et al (2009) and aims to determine the prevalence and persistence of postpartum physical symptoms (Chien et al, 2009). The Turkish validity and reliability study of the scale was carried out by Arkan (2016). In the study of Arkan (2016), the internal consistency of the scale was determined to be at a very reliable level (Cronbach α=0.79). In this study, the cronbach α value of the scale will be calculated.
  The scale consists of 18 items. Each item of the scale is in a 4-point Likert format and these items are evaluated as 0 (absent), 1 (mild), 2 (moderate), and 3 (high). Scale total score ranges from 0 to 54. High scores obtained from the scale indicate that the severity of postpartum physical symptoms is high (Arkan, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Gülten Koç, Study Director — Hacettepe University
Locations (1):
- University of Health Sciences Etlik Zübeyde Hanim Gyn Diseases Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, CSR
Time Frame: march, 2022
Access Criteria: When the study is converted into a protocol or an article, it will be published in an international journal by the researchers.

REFERENCES:
- [Derived] Oztoprak PU, Koc G, Erkaya S. Evaluation of the effect of a nurse navigation program developed for postpartum mothers on maternal health: A randomized controlled study. Public Health Nurs. 2023 Sep-Oct;40(5):672-684. doi: 10.1111/phn.13226. Epub 2023 Jul 13. PMID 37443414